CLINICAL TRIAL: NCT06179667
Title: Gulhane Training and Research Hospital
Brief Title: Development and Effectiveness of a User-centered Mobile Application for Informal Caregivers of People Living With Dementia: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Buğse Yüceer, Phd Student, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: --De-Mobile--001
Record Dates: First submitted 2023-11-27; First posted 2023-12-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Dementia
Keywords: Dementia; Informal caregiver; Mobile application; Care burden; Quality of life; Neuropsychiatric symptom
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Caregivers will be encouraged to use the mobile application every day during the implementation period of the study (two months).
  Interventions: Behavioral: Mobile Application
- Control Group (No Intervention): No treatment will be performed on individuals in the control group.

INTERVENTIONS:
Behavioral: Mobile Application — It is aimed to develop the mobile application to address the problems and training needs of informal caregivers regarding the caregiving process. In this context, in order to determine the needs of caregivers, face-to-face in-depth interviews will be held with caregivers using the "Semi-Structured Questionnaire for Qualitative Interviews" at the University of Health Sciences GTRH Geriatrics Department. The content of the mobile application will be created according to the topics determined as a result of qualitative research. Technical development of the application will be carried out by the web application designer.
  Arms: Intervention Group

SUMMARY:
The research shows that the mobile application developed for informal caregivers of people living with dementia affects caregivers' care burden, quality of life; It was planned as a mixed-type, randomized controlled study to evaluate its effect on the neuropsychiatric symptoms of individuals with dementia. The research is planned to be conducted at the Geriatrics Department of Gülhane Training and Research Hospital (GTRH) between August 2023 and December 2025.The population of the research consists of informal caregivers of people living with dementia who are followed up in the Geriatrics department. As a result of the power analysis performed in the G-power 3.1.9.4 package program based on the reference article, it was calculated that the sample size should be 74 in total, 37 caregivers for each group. Considering the 15% data loss rate, the sample size was determined as 86 in total, 43 caregivers for each group.t is aimed to develop the mobile application to address the problems and training needs of informal caregivers regarding the caregiving process. In this context, in order to determine the needs of caregivers, face-to-face in-depth interviews will be held with caregivers using the "Semi-Structured Questionnaire for Qualitative Interviews" at the University of Health Sciences GTRH Geriatrics Department. The content of the mobile application will be created according to the topics determined as a result of qualitative research. Examining the Effectiveness of the Developed Mobile Application Individuals who meet the inclusion criteria and agree to participate in the study will be assigned to the intervention and control groups by simple randomization method.Caregivers in intervention group will be encouraged to use the mobile application every day during the implementation of the research (two months). No treatment will be performed on individuals in the control group. At the end of the research (2nd month), data will be collected electronically through a survey using the Zarit Care Burden Scale, WHOQOL, Neuropsychiatric Inventory.

DETAILED DESCRIPTION:
Due to the decrease in cognitive functions in individuals with dementia, individuals experience difficulties in performing daily living activities. In the later stages of dementia, behavioral symptoms such as personality changes, hallucinations, and agitation are also observed. All these cognitive, functional and behavioral symptoms that occur due to dementia cause the degree of addiction of the individual with dementia to increase. Care of individuals with dementia is generally provided by informal caregivers, including friends, neighbors, and family members. The responsibilities undertaken by individuals providing informal care during the dementia process cause individuals to be affected socially, physically and economically. All these problems cause care burden on caregivers, leading to a decrease in their quality of life and involuntary treatment of individuals with dementia, resulting in more neuropsychiatric syndromes in individuals. In this context, caregivers need to be supported with practices that will enable them to cope effectively with the caregiving process. There are non-pharmacological practices such as psychotherapy, support groups, meditation/mindfulness in the literature to support informal caregivers. However, since these applications occur within a certain period of time, their effects do not last long . Caregivers need resources that have a long-lasting effect and that they can benefit from when they need them. In this context, mobile applications are used in the literature. Mobile applications are very advantageous applications in terms of cost and time effectiveness that can enable personalized training opportunities and can be carried with the person 24 hours a day. There are a limited number of mobile applications in the literature developed for comprehensive support of informal caregivers.For this reason, this research is planned to examine the effectiveness of the mobile application developed for informal caregivers of individuals with dementia.

Place and Time of Research The research is planned to be conducted at the Geriatrics Polyclinic of Gülhane Training and Research Hospital between August 2023 and December 2025.

Population and Sample of the Research:

The population of the research consists of informal caregivers of people living with dementia who are followed up in the Geriatrics outpatient clinic of Health Sciences University GTRH. As a result of the power analysis performed in the G-power 3.1.9.4 package program based on the reference article, it was calculated that the sample size should be 74 in total, 37 caregivers for each group. Considering the 15% data loss rate, the sample size was determined as 86 in total, 43 caregivers for each group.

Research Inclusion Criteria:

* Being over 18 years old
* Reading/writing Turkish
* Being an informal caregiver of an individual diagnosed with Major Neurodegenerative Disorders (dementia) by a physician according to DSM 5 criteria
* Providing care to the individual with dementia for at least 6 hours a day for at least 1 month
* No neurological or psychiatric problems
* Having a smart phone with internet connection and being able to use the application program

Criteria for Exclusion from the Research:

* Being a formal caregiver of an individual diagnosed with Major Neurodegenerative Disorders (dementia) by a physician according to DSM 5 criteria
* Failure to log into the mobile application at least once a week during the study period (two months) Data Collection Tools
* Form Regarding Sociodemographic and Caregiving Characteristics of Caregivers
* Zarit Care Burden Scale
* World Health Organization Quality of Life Scale Short Form (WHOQOL)
* Neuropsychiatric Inventory (NPE)
* Semi-Structured Questionnaire for Qualitative Interviews
* Quality Criteria for Consumer Health Information (DISCERN) Scale
* Mobile Application Usability Scale
* System Usability Scale Data Collection and Application Stage 1: Development of Mobile Application It is aimed to develop the mobile application to address the problems and training needs of informal caregivers regarding the caregiving process. In this context, in order to determine the needs of caregivers, face-to-face in-depth interviews will be held with caregivers using the "Semi-Structured Questionnaire for Qualitative Interviews" at the University of Health Sciences GTRH Geriatrics Department. The content of the mobile application will be created according to the topics determined as a result of qualitative research. Technical development of the application will be carried out by the web application designer. The mobile application will be presented to expert academicians using the DISCERN scale and the Mobile Application Usability Scale to be evaluated in terms of the suitability and usability of its content.

Stage 2: Examining the Effectiveness of the Developed Mobile Application Individuals who meet the inclusion criteria and agree to participate in the study will be assigned to the intervention and control groups by simple randomization method.

- During the first interview, the consent of individuals in the intervention and control groups will be obtained and information about the research process will be given. Data were collected online using the Informal Caregivers' Sociodemographic and Caregiving Characteristics Form, the Zarit Care Burden Scale, WHOQOL, NPE.

Intervention Group;

* Caregivers will be encouraged to use the mobile application every day during the implementation of the research (two months).
* At the end of the application (2nd month), Zarit Care Burden Scale, WHOQOL, NPE; System Usability Scale. Data will be collected electronically.

Control Group;

* No treatment will be performed on individuals in the control group.
* At the end of the research (2nd month), data will be collected electronically through a survey using the Zarit Care Burden Scale, WHOQOL, Neuropsychiatric Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Reading/writing Turkish
* Being an informal caregiver of an individual diagnosed with Major Neurodegenerative Disorders (dementia) by a physician according to DSM 5 criteria
* Providing care to the individual with dementia for at least 6 hours a day for at least 1 month
* No neurological or psychiatric problems
* Having a smart phone with internet connection and being able to use the application program

Exclusion Criteria:

* Being a formal caregiver of an individual diagnosed with dementia by a physician according to DSM 5 criteria
* During the two-month application period of the study, I did not log into the mobile application at least once a week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
caregivers' care burden scores, quality of life scores and neuropsychiatric inventory scores | At the end of the intervention (2nd month)
  Change of caregivers' care burden scores, quality of life scores and neuropsychiatric inventory scores

CONTACTS AND LOCATIONS:
Locations (1):
- Gülhane Research and Training Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No